CLINICAL TRIAL: NCT01262027
Title: A Phase II Study of TKI258 (Dovitinib Lactate) as Salvage Therapy in Patients With Stage IV HER2-negative Inflammatory Breast Cancer (IBC) and Local or Distant Relapse
Brief Title: TKI258 for Metastatic Inflammatory Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0296; NCI-2011-00299 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Metastatic inflammatory breast cancer; Stage IV disease; HER2-negative; Dovitinib; TKI258
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Disease | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dovitinib (Experimental): A complete treatment cycle defined as 28 days or 4 weeks (+/- 2 days). Patients receive a single daily oral dose of 500 mg of dovitinib for 5 consecutive days, followed by a 2-day rest period (5 days on/2 days off schedule).
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — 500 mg by mouth for 5 consecutive days, followed by a 2-day rest period (5 days on/2 days off schedule) for every 28 day cycle.
  Other Names: TKI258

SUMMARY:
The goal of this clinical research study is to learn if dovitinib can help to control inflammatory breast cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Dovitinib is designed bind to a protein on the surface of cancer cells called the FGF receptor. This may slow the growth of cancer cells or kill cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take dovitinib by mouth each day for 5 days and have a 2-day rest period (5 days on/2 days off schedule). The first dose of each week is Day 1. You should take dovitinib in the morning with a glass (about 8 ounces) of water at least 1 hour before or at least 2 hours after eating. It is important that you take the study drug at about the same time every day.

If you forget to take a dose of the study drug as scheduled, or take a dose during your 2-day rest period, you should follow the guidelines below or call your study staff:

* If you take a dose on Day 6, then you will rest on Day 7 and start taking the drug on Day 1.
* If you take a dose on Day 7, then you will skip Day 1 the next schedule and start dosing on Day 2.
* If you take a dose on Day 6 and Day 7, then you will skip Days 1 and 2 of the next schedule and start dosing on Day 3.
* If you missed a dose on Days 1, 2, 3, or 4, you should restart the next dosing day and rest on Days 6 and 7.
* If you missed a dose on Day 5, you should rest on Days 6 and 7, and restart dosing on Day 1 of the next week.

You should not take additional medications including over-the-counter products and herbal/alternative medications during the study without asking your doctor. It is important to avoid medications that are known to cause liver side effects.

If you experience intolerable side effects, the study doctor may give you drugs to help control the side effects.

You should store the study drug at room temperature and out of direct sunlight. The study drug should also be kept away from children.

About every 4 weeks, you will need to bring back your empty or partially used bottles of study drug.

During Treatment:

At every visit, you will be asked if you have had any side effects.

Before each Cycle:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Cycle 1, around Days 8 and 22:

° Blood (about 1 tablespoon) will be drawn to check your liver function.

Cycle 2 around Day 8:

° Blood (about 1 tablespoon) will be drawn to check your liver function.

Every 2 cycles (before Cycles 3, 5, 7, and so on):

* If the doctor thinks it is needed, photographs will be taken of your skin and any areas affected by inflammatory breast cancer.
* If the doctor thinks it is needed, you will have x-rays, a CT scan of the chest and/or abdomen, and/or a bone scan.

Before Cycle 3:

* If the doctor thinks it is needed, you will have a positron emission computed tomography (PET/CT) scan to check the status of the disease.
* Blood (about 2 tablespoons) will be drawn for biomarker testing.

You will also have a one-time blood draw (about 1 tablespoon) to measure the level of the study drug in your blood. This sample may be drawn on Days 12 or 26 of Cycle 1, before Cycle 2, or on Day 12 of Cycle 2.

If the doctor thinks it is needed, any of these tests and procedures may be performed earlier. If the doctor thinks it is needed, you will have an ECG, ECHO, or MUGA scan to check your heart function.

Length of Study:

You may remain on study for as long as you are benefiting. You will be taken off study treatment if the disease gets worse or you experience intolerable side effects.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End-of-Treatment Visit:

After you are off study, you will have a end-of-treatment visit within 14 days after the last study visit.

* You will be asked if you have had any side effects.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, photographs will be taken of your skin and any areas affected by inflammatory breast cancer.
* If the doctor thinks it is needed, you will have x-rays, a CT scan of the chest and/or abdomen, and/or a bone scan.
* If the doctor thinks it is needed, you will have an ECG and ECHO or MUGA scan to check your heart function.
* If the doctor thinks it is needed, you will have a PET/CT scan to check the status of the disease.

Follow-up Visits:

You will be called or e-mailed every 3 months for up to 1 year and asked how you are doing.

This is an investigational study. Dovitinib is not FDA approved or commercially available. At this time, dovitinib is only being used in research.

Up to 33 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have histological confirmation of breast carcinoma with a clinical diagnosis of IBC based on presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d orange), with or without an underlying palpable mass involving the majority of the skin of the breast. Pathological evidence of dermal lymphatic invasion should be noted but is not required for diagnosis.
2. Patients have stage IV disease with local or distant relapse
3. Patients have negative HER2 expression by IHC (defined as 0 or1+), or fluorescence in situ hybridization (FISH). If HER2 is 2+, negative HER2 expression must be confirmed by FISH.
4. Patients are able to swallow and retain oral medication.
5. Patients have Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Patients have received two or more standard chemotherapies for metastatic disease and have relapsed.
7. Patients have ability and willingness to sign written informed consent.
8. Patients are 18 years of age or older.
9. Female patients of childbearing potential (A female not free from menses > 2 years or not surgically sterilized) must be willing to use highly effective contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study. Highly effective contraception, defined as male condom with spermicide, diaphragm with spermicide, intra-uterine device. Highly effective contraception must be used by both sexes during the study and must be continued for 8 weeks after the end of study treatment. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
10. Female patients of childbearing potential must have negative serum pregnancy test </=14 days prior to starting study treatment.
11. If Patients have been treated with anti-vascular endothelial growth factor (VEGF) agents, such as Bevacizumab, last dose must be > 4 weeks.
12. Patients have biopsy tissue of the metastatic disease (including chest wall or regional nodes) available (paraffin blocks or up to 20 unstained slides), if no biopsy tissue available, a biopsy (or thoracentesis if patient has pleural effusion only) of the metastatic disease will be performed to confirm the diagnoses.
13. Serum total bilirubin must be within Upper Limited Normal (T. Bilirubin upper limit of normal (ULN)=1.0 mg/dl)
14. AST and ALT must be < 2.5 x ULN(with or without liver metastases).

Exclusion Criteria:

1. Patients are receiving concurrent anti-cancer therapy (chemotherapy, immunotherapy, radiation therapy and biological therapy) while taking study medication.
2. Cirrhosis of liver, or known hepatitis B or C infection have hepatic impairment Child-Pugh Score of B or worse.
3. Absolute neutrophil count (ANC) < 1.5
4. Patients have an active infection and require IV or oral antibiotics.
5. Impaired cardiac function or clinically significant cardiac diseases, including any of the following: a) History or presence of serious uncontrolled ventricular arrhythmias or presence of atrial fibrillation; b) Clinically significant resting bradycardia (< 50 beats per minute); c) left ventricular ejection fraction (LVEF) assessed by 2-D echocardiogram (ECHO) < 50% or lower limit of normal (which ever is higher) or multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (which ever is higher). d) Any of the following within 6 months prior to study entry: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE); e) Uncontrolled hypertension defined by an SBP>150 and/or a diastolic blood pressure (DBP)>100 mm Hg with or without anti-hypertensive medication.
6. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
7. Patients have a concurrent disease or condition that would make them inappropriate for study participation, or any serious medical disorder that would interfere with patients safety.
8. Patients with only locally or regionally confined disease without evidence of metastatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 27, 2012 to July 29, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Dovitinib: Dovitinib 500 mg single oral dose for 5 consecutive days, followed by a 2-day rest period (5 days on/2 days off schedule) for every 28 day cycle.
Period: Overall Study
Arm/Group | Dovitinib
Started | 22
Completed | 17
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dovitinib
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Complete Response [CR], Partial Response [PR] or Stable Disease [SD]) of Participants
Description: Number of participants experiencing CR, PR or SD as defined by Response Evaluation Criteria In Solid Tumors (RECIST). Response is anyone who experiences SD, CR or PR in first 6 months. CR: Disappearance clinical evidence active tumor by evaluation, mammogram & ultrasound. No symptoms or evidence of residual invasive tumor, including no residual tumor in axillary lymph nodes. PR: 50%/> decrease for minimum 4 weeks in measurable lesion determined by product of perpendicular diameters of lesion. Every lesion should not regress to qualify as PR; however, if lesion progresses or if new lesions appear, response cannot be classified as PR. Minor Response [MR]: Decreases in tumor masses insufficient to qualify as partial remission, i.e. <50%. SD: Between MR & PD. PD: Increase 25% measured lesion from baseline. New lesions constitutes increasing disease. Mixed responses consid
Time Frame: 6 months
Population: Three participants were not evaluable for response due to early departure from study.
Measure: Number; unit: participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 19
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 1

2. Secondary Outcome: Safety Analysis of Dovitinib: Most Frequently Reported Treatment-related Adverse Event (AEs)
Description: Safety analysis evaluated by grading each adverse event according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and reporting the type, frequency and severity in a summary format. Full AE reporting can be found in the Adverse Event Section.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 22
Participants
  Grade 3 & 4: Fatigue | 5
  Grade 3 & 4: Pain | 3

ADVERSE EVENTS:
Time Frame: Adverse event collection was from for a complete treatment cycle defined as 28 days or 4 weeks (+/- 2 days) up to six cycles (24 weeks) and/or up to 30 days following discontinuation of study drug.
Arm/Group | Dovitinib
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=22)
Blood bilirubin increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=22)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1)
Chest wall pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dyspnea (Gastrointestinal disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Ejection fraction decreased (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 11 (17)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - Sinus (Infections and infestations) | 2 (2)
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 12 (12)
Neck pain (General disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT01262027/Prot_SAP_000.pdf